CLINICAL TRIAL: NCT05174689
Title: Epigenetic Regulation of Excercise Induced Asthma
Brief Title: Epigenetic Regulation of Exercise Induced Asthma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Stefan Zielen, Prof. Dr. med., Johann Wolfgang Goethe University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: E68/21
Record Dates: First submitted 2021-08-30; First posted 2022-01-03 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Exercise Induced Asthma; House Dust Mite Allergy
Keywords: Exercise Induced Asthma; eNO; exercise challenge; micro RNAs
MeSH Terms: conditions — Asthma, Exercise-Induced; Dust Mite Allergy

STUDY DESIGN:
Intervention Model Description: The micro RNA profile of patients with known EIA and house dust mite allergy and patients with EIA without allergic sensitization are compared to the micro RNA profile of healthy controls
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EIA wih house dust mite (Other): Patients with EIA and house-dust mite allergy and an eNO > 30 ppb
  Interventions: Diagnostic Test: Exercise challenge in the cold chamber (ECC); Diagnostic Test: mRNA profile; Diagnostic Test: standard diagnostic
- EIA without sensitization (Other): Patients with EIA without allergic sensitization and an eNO < 20 ppb
  Interventions: Diagnostic Test: Exercise challenge in the cold chamber (ECC); Diagnostic Test: mRNA profile; Diagnostic Test: standard diagnostic
- Healthy controls (Other): Healthy controls without allergic sensitization or known asthma
  Interventions: Diagnostic Test: mRNA profile; Diagnostic Test: standard diagnostic

INTERVENTIONS:
Diagnostic Test: Exercise challenge in the cold chamber (ECC) — Exercise challenge (defined as running on a treadmill for 6-8 minutes on submaximal work load in a cold chamber. Gradient: 10%, temperature 2-4°C. After the exercise challenge controlling bodyplethysmography and spirometry after 5, 10, 15 and 30 minutes. A positive reaction is a decrease of ≥ 10% of FEV1 in comparison to the initial value.
  Arms: EIA wih house dust mite; EIA without sensitization
Diagnostic Test: mRNA profile — Blood taking with full blood exam and PAXgene tube for investigation oft the micro RNA profiles. The PAXgene Blood RNA kit insulates total RNA inclusive miRNA and small RNA which are centrifugated, pelletised, washed and incubated to detach proteins. For mapping the particular miRNA there will be generated libraries with specifical codes to match the analysis to the original probe. Next generation sequencing will be performed by MISeq REagent Kit v3 and the analysis oft the different expressions in the R Version 3.2.3. The divergent expressions will be refurbished by computer and databased.
Diagnostic Test: standard diagnostic — bodyplethysmography, spirometry, exhaled NO, skin prick test, asthma control test (ACT)

SUMMARY:
The purpose of this study is to investigate the micro ribonucleic acid (mRNA) profiles of patients with EIA without allergic sensitization and EIA with house dust mite sensitization compared to that of healthy controls.

DETAILED DESCRIPTION:
Patients with known EIA are periodically reexamined by medical history, clinical examination, bodyplethysmography, spirometry, exhaled nitric oxide (eNO), skin prick test, methacholin challenge test and exercise-challenge in a cold-chamber at 2-4°C (ECC). Additionally the investigators gathers the questionnaires: Asthma Control Test (ACT) and Dyspnoe Index (DI).

Besides these standard procedures the investigators want to investigate the micro-RNA profiles in two EIA subgroups: EIA with house-dust allergy (n = 24) and EIA without house-dust allergy (n = 24).

Both groups are characterized by different eNO levels. The patients with EIA and house-dust allergy should have an eNO > 30 ppb, the patients with EIA without house-dust allergy an eNO < 20 ppb.

The micro-RNA profiles of the both EIA subgroups will be compared the micro RNA profiles of 20 healthy controls .

Therefore blood will be taken (for a complete blood count and micro RNA analysis) at three points of time: before ECC, directly after ECC and after 24 hours ± 4 hours after ECC.

ELIGIBILITY:
For EIA patients

Inclusion Criteria:

* written agreement
* age >=12 and <= 24
* known exercise induced asthma
* Group 1: skin prick test positiv house-dust allergy, eNO > 30 ppb, MCT PD20 < 0,1 mg
* Group 2: skin prick test negative house-dust allergy, eNO < 20 ppb, MCT PD20 < 1 mg
* lung function before ECC forced vital capacity (FVC) ≥ 75% and forced exspiratory pressure in one second (FEV1) ≥ 70%

Exclusion Criteria:

* age < 12 und > 24 years
* lung function FVC < 75% und FEV1< 70%
* inability to understand the range of the study
* chronic asthma with systemic cortisone therapy
* regular therapy with inhalative corticosteroids or leukotriene-antagonists <14 days before visit 1
* intake of long acting beta-agonists (LABA) 48 h before examination
* intake of short acting beta-agonists (SABA) 8 h before examination
* acute severe infection (pneumonia) within the last 4 weeks
* other chronic diseases or infections (HIV, Tbc)
* pregnancy

For healthy controls

Inclusion Criteria:

* written agreement
* age >=18 and <= 24

Exclusion Criteria:

* age < 18 and > 24 years
* known asthma bronchiale or other chronic lung diseases
* lung function FVC < 90% and FEV1 < 80%
* allergic sensitization in skin prick test
* eNO > 30 ppb
* inability to understand the range of the study
* acute severe infection (pneumonia) within the last 4 weeks
* other chronic diseases or infections (HIV, Tbc)
* pregnancy

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 68 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Dysregulation of miRNA-146 | 1 Year
  The primary endpoint is the dysregulation of miRNA-146 in comparison to the control group and within the subgroups which play an determined role in the bronchial inflammation.
  Therefore the total RNA, including miRNA, will be isolated using the PAXgene Blood miRNA Kit (Qiagen, Hilden, Germany). Concentration of RNA will be assessed using Nanodrop Lite spectrometry (Thermo Scientific, Dreieich, Germany). MiRNA libraries are generated with the QIAseq miRNA Library Kit (Qiagen, Hilden, Germany). Next generation sequencing (NGS) will be performed with the MiSeq Reagent Kit v3, the PhiX Sequencing Control v3 and the MiSeq™ Desktop Sequencer (all Illumina Inc., San Diego, CA, USA). Differential expression analysis will be performed in RStudio 1.2.1335 (https://cran.r-project.org/). False discovery rate correction will be applied and miRNAs are considered to be differentially expressed with p < 0.05.

SECONDARY OUTCOMES:
Dysregulation miRNAs affecting Th2 mediated bronchial inflammation (miRNA-126, miRNA-21, miRNA-145, let7-mimic) | 1 Year
  Dysregulation of other miRNAs affecting the Th2 mediated bronchial inflammation (miRNA-126, miRNA-21, miRNA-145, let7-mimic) and compare to the control group.
  MiRNA preparation and measurement processes are described in Outcome 1.
Cange of eNO | 1 Year
  Change of eNO after ECC in the EIA subgroups compared to the healthy controls
Change of leucocytes and neutrophile granulocytes | 1 Year
  Change of leucocytes and neutrophile granulocytes after ECC in the EIA subgroups compared to the healthy controls
FEV1-decrease in ECC | 1 Year
  Comparison of the FEV1-decrease in ECC with significant dysregulated miRNA in the EIA subgroups compared to the healthy controls
Comparison eNO with significant dysregulated miRNA | 1 Year
  Comparison of the initial value of exhaled NO with significant dysregulated miRNA in the EIA subgroups compared to the healthy controls
Comparison of change of leucocytes and neutrophile granulocytes with significant dysregulated miRNA | 1 Year
  Comparison of the increase of leucocytes and neutrophile granulocytes after ECC significant dysregulated miRNA in the EIA subgroups compared to the healthy controls
Comparison of ACT with significant dysregulated miRNA | 1 Year
  Comparison of the score in ACT with significant dysregulated miRNA in the EIA subgroups compared to the healthy controls
Comparison of DI with significant dysregulated miRNA | 1 Year
  Comparison of the scoresin DI with significant dysregulated miRNA in the EIA subgroups compared to the healthy controls

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Dreßler, MD, Principal Investigator — Johann Wolfgang Goethe University Hospital
Locations (1):
- Universitätsklinikum Frankfurt, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parsons JP, Hallstrand TS, Mastronarde JG, Kaminsky DA, Rundell KW, Hull JH, Storms WW, Weiler JM, Cheek FM, Wilson KC, Anderson SD; American Thoracic Society Subcommittee on Exercise-induced Bronchoconstriction. An official American Thoracic Society clinical practice guideline: exercise-induced bronchoconstriction. Am J Respir Crit Care Med. 2013 May 1;187(9):1016-27. doi: 10.1164/rccm.201303-0437ST. PMID 23634861
- [Background] Dressler M, Friedrich T, Lasowski N, Herrmann E, Zielen S, Schulze J. Predictors and reproducibility of exercise-induced bronchoconstriction in cold air. BMC Pulm Med. 2019 May 16;19(1):94. doi: 10.1186/s12890-019-0845-3. PMID 31097027
- [Background] Dressler M, Salzmann-Manrique E, Zielen S, Schulze J. Exhaled NO as a predictor of exercise-induced asthma in cold air. Nitric Oxide. 2018 Jun 1;76:45-52. doi: 10.1016/j.niox.2018.03.004. Epub 2018 Mar 8. PMID 29526567
- [Background] Schulze J, Smith HJ, Fuchs J, Herrmann E, Dressler M, Rose MA, Zielen S. Methacholine challenge in young children as evaluated by spirometry and impulse oscillometry. Respir Med. 2012 May;106(5):627-34. doi: 10.1016/j.rmed.2012.01.007. Epub 2012 Feb 10. PMID 22326606
- [Background] Schulze J, Rosewich M, Riemer C, Dressler M, Rose MA, Zielen S. Methacholine challenge--comparison of an ATS protocol to a new rapid single concentration technique. Respir Med. 2009 Dec;103(12):1898-903. doi: 10.1016/j.rmed.2009.06.007. Epub 2009 Jul 10. PMID 19596563
- [Background] Schulze J, Rosewich M, Dressler M, Riemer C, Rose MA, Zielen S. Bronchial allergen challenge using the Medicaid dosimeter. Int Arch Allergy Immunol. 2012;157(1):89-97. doi: 10.1159/000324473. Epub 2011 Sep 7. PMID 21912178
- [Background] Schulze J, Voss S, Zissler U, Rose MA, Zielen S, Schubert R. Airway responses and inflammation in subjects with asthma after four days of repeated high-single-dose allergen challenge. Respir Res. 2012 Sep 19;13(1):78. doi: 10.1186/1465-9921-13-78. PMID 22989372
- [Background] Anderson SD, Charlton B, Weiler JM, Nichols S, Spector SL, Pearlman DS; A305 Study Group. Comparison of mannitol and methacholine to predict exercise-induced bronchoconstriction and a clinical diagnosis of asthma. Respir Res. 2009 Jan 23;10(1):4. doi: 10.1186/1465-9921-10-4. PMID 19161635
- [Background] Driessen JM, van der Palen J, van Aalderen WM, de Jongh FH, Thio BJ. Inspiratory airflow limitation after exercise challenge in cold air in asthmatic children. Respir Med. 2012 Oct;106(10):1362-8. doi: 10.1016/j.rmed.2012.06.017. Epub 2012 Jul 11. PMID 22789953
- [Background] Zielen S, Lieb A, De La Motte S, Wagner F, de Monchy J, Fuhr R, Munzu C, Koehne-Voss S, Riviere GJ, Kaiser G, Erpenbeck VJ. Omalizumab protects against allergen- induced bronchoconstriction in allergic (immunoglobulin E-mediated) asthma. Int Arch Allergy Immunol. 2013;160(1):102-10. doi: 10.1159/000339243. Epub 2012 Aug 28. PMID 22948442
- [Background] Rosewich M, Zissler UM, Kheiri T, Voss S, Eickmeier O, Schulze J, Herrmann E, Ducker RP, Schubert R, Zielen S. Airway inflammation in children and adolescents with bronchiolitis obliterans. Cytokine. 2015 May;73(1):156-62. doi: 10.1016/j.cyto.2014.10.026. Epub 2015 Mar 6. PMID 25748838
- [Background] Jerkic SP, Michel F, Donath H, Herrmann E, Schubert R, Rosewich M, Zielen S. Calprotectin as a New Sensitive Marker of Neutrophilic Inflammation in Patients with Bronchiolitis Obliterans. Mediators Inflamm. 2020 May 1;2020:4641585. doi: 10.1155/2020/4641585. eCollection 2020. PMID 32410855
- [Background] Fussbroich D, Kohnle C, Schwenger T, Driessler C, Ducker RP, Eickmeier O, Gottwald G, Jerkic SP, Zielen S, Kreyenberg H, Beermann C, Chiocchetti AG, Schubert R. A combination of LCPUFAs regulates the expression of miRNA-146a-5p in a murine asthma model and human alveolar cells. Prostaglandins Other Lipid Mediat. 2020 Apr;147:106378. doi: 10.1016/j.prostaglandins.2019.106378. Epub 2019 Nov 4. PMID 31698144
- [Background] Tan Z, Randall G, Fan J, Camoretti-Mercado B, Brockman-Schneider R, Pan L, Solway J, Gern JE, Lemanske RF, Nicolae D, Ober C. Allele-specific targeting of microRNAs to HLA-G and risk of asthma. Am J Hum Genet. 2007 Oct;81(4):829-34. doi: 10.1086/521200. Epub 2007 Aug 20. PMID 17847008
- [Background] Zhang YY, Zhong M, Zhang MY, Lv K. [Expression and clinical significance of miR-155 in peripheral blood CD4(+);T cells of patients with allergic asthma]. Xi Bao Yu Fen Zi Mian Yi Xue Za Zhi. 2012 May;28(5):540-3. Chinese. PMID 22558995
- [Background] Lu TX, Munitz A, Rothenberg ME. MicroRNA-21 is up-regulated in allergic airway inflammation and regulates IL-12p35 expression. J Immunol. 2009 Apr 15;182(8):4994-5002. doi: 10.4049/jimmunol.0803560. PMID 19342679
- [Background] Mattes J, Collison A, Plank M, Phipps S, Foster PS. Antagonism of microRNA-126 suppresses the effector function of TH2 cells and the development of allergic airways disease. Proc Natl Acad Sci U S A. 2009 Nov 3;106(44):18704-9. doi: 10.1073/pnas.0905063106. Epub 2009 Oct 20. PMID 19843690
- [Background] Williams AE, Larner-Svensson H, Perry MM, Campbell GA, Herrick SE, Adcock IM, Erjefalt JS, Chung KF, Lindsay MA. MicroRNA expression profiling in mild asthmatic human airways and effect of corticosteroid therapy. PLoS One. 2009 Jun 12;4(6):e5889. doi: 10.1371/journal.pone.0005889. PMID 19521514
- [Background] Polikepahad S, Knight JM, Naghavi AO, Oplt T, Creighton CJ, Shaw C, Benham AL, Kim J, Soibam B, Harris RA, Coarfa C, Zariff A, Milosavljevic A, Batts LM, Kheradmand F, Gunaratne PH, Corry DB. Proinflammatory role for let-7 microRNAS in experimental asthma. J Biol Chem. 2010 Sep 24;285(39):30139-49. doi: 10.1074/jbc.M110.145698. Epub 2010 Jul 14. PMID 20630862
- [Background] Chiba Y, Tanabe M, Goto K, Sakai H, Misawa M. Down-regulation of miR-133a contributes to up-regulation of Rhoa in bronchial smooth muscle cells. Am J Respir Crit Care Med. 2009 Oct 15;180(8):713-9. doi: 10.1164/rccm.200903-0325OC. Epub 2009 Jul 30. PMID 19644046
- [Background] Kumar M, Mabalirajan U, Agrawal A, Ghosh B. Proinflammatory role of let-7 miRNAs in experimental asthma? J Biol Chem. 2010 Nov 26;285(48):le19: author reply le20. doi: 10.1074/jbc.L110.145698. No abstract available. PMID 21097512
- [Background] Garbacki N, Di Valentin E, Huynh-Thu VA, Geurts P, Irrthum A, Crahay C, Arnould T, Deroanne C, Piette J, Cataldo D, Colige A. MicroRNAs profiling in murine models of acute and chronic asthma: a relationship with mRNAs targets. PLoS One. 2011 Jan 28;6(1):e16509. doi: 10.1371/journal.pone.0016509. PMID 21305051
- [Background] Mayoral RJ, Pipkin ME, Pachkov M, van Nimwegen E, Rao A, Monticelli S. MicroRNA-221-222 regulate the cell cycle in mast cells. J Immunol. 2009 Jan 1;182(1):433-45. doi: 10.4049/jimmunol.182.1.433. PMID 19109175
- [Background] Liu X, Nelson A, Wang X, Kanaji N, Kim M, Sato T, Nakanishi M, Li Y, Sun J, Michalski J, Patil A, Basma H, Rennard SI. MicroRNA-146a modulates human bronchial epithelial cell survival in response to the cytokine-induced apoptosis. Biochem Biophys Res Commun. 2009 Feb 27;380(1):177-82. doi: 10.1016/j.bbrc.2009.01.066. Epub 2009 Jan 22. PMID 19167348
- [Background] Sharma A, Kumar M, Ahmad T, Mabalirajan U, Aich J, Agrawal A, Ghosh B. Antagonism of mmu-mir-106a attenuates asthma features in allergic murine model. J Appl Physiol (1985). 2012 Aug;113(3):459-64. doi: 10.1152/japplphysiol.00001.2012. Epub 2012 Jun 14. PMID 22700801
- [Background] Feng MJ, Shi F, Qiu C, Peng WK. MicroRNA-181a, -146a and -146b in spleen CD4+ T lymphocytes play proinflammatory roles in a murine model of asthma. Int Immunopharmacol. 2012 Jul;13(3):347-53. doi: 10.1016/j.intimp.2012.05.001. Epub 2012 May 10. PMID 22580216
- [Background] Omran A, Elimam D, Yin F. MicroRNAs: new insights into chronic childhood diseases. Biomed Res Int. 2013;2013:291826. doi: 10.1155/2013/291826. Epub 2013 Jun 27. PMID 23878802